CLINICAL TRIAL: NCT03225534
Title: Project 500 CHILD Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Collaborators: Allergy, Genes and Environment Network (AllerGen) NCE (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); St. Joseph's Healthcare Hamilton (Other); University of Toronto (Other); University of Manitoba (Other); University of Alberta (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Malcolm Sears, Professor of Medicine, McMaster University
Other Study IDs: Project 500 ISS
Record Dates: First submitted 2017-07-07; First posted 2017-07-21 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Asthma in Children; Allergy in Children; Environmental Exposure; Genetic Predisposition
Keywords: Asthma; Allergy; Epidemiology; Environment; Exposures
MeSH Terms: conditions — Genetic Predisposition to Disease; Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cord blood. Child 1 year blood Child 5 year blood. Parental venous blood. Saliva samples. Urine samples. Stool samples. Breast milk samples. Nasal swabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This proposal relates to the testing of several specific hypotheses in a subset of 500 participants in the Canadian Healthy Infant Longitudinal Development (CHILD) Study. These 500 now have complete data from the time of recruitment (in pregnancy) to age 1 year. The primary purpose of this proposal is to identify risk factors for early allergic outcomes and biomarkers that may predict future disease. These 500 infants will provide critical preliminary data, not only related to early outcomes, but also to inform analytical plans for the full CHILD cohort.

DETAILED DESCRIPTION:
The objective of Project 500 is to carefully analyze a complete set of multiple clinical and environmental questionnaires and selected infant biological samples pertinent to early clinical outcomes (up to age 1 year). The primary clinical outcomes are recurrent episodes of wheezing and development of atopy by age 1 year. Atopy is defined by skin allergen responses. Secondary outcomes include atopic dermatitis or eczema, and reported food allergy. The investigators propose detailed exploration of patterns of clinical illnesses and will correlate these with analysis of multiple biomarkers to determine their predictive power.

There is good evidence from longitudinal epidemiological studies and from clinical trials that allergy is both a common precursor to childhood asthma and also a predictor of persistence of childhood asthma into adulthood. The "atopic march" is a well recognized phenomenon in which children develop atopic dermatitis and/or food allergy in early childhood, and then go on to have recurrent wheezing and persistent atopic asthma in later childhood and adulthood. The selection of specific hypotheses for examination in Project 500 reflects this phenomenon.

Four specific hypotheses will be tested in "Project 500":

1. Maternal diet in pregnancy influences food sensitization in infancy; specifically avoidance of foods (e.g. peanuts) is associated with intolerance to that food.

   Research on diet and interventions to prevent atopic disease have focused on foods with anti-inflammatory properties (e.g. n-3 fatty acids), antioxidants (vitamin E and zinc), and vitamin D. Recent meta-analyses suggest beneficial effects for pre-natal vitamins A, D, and E, zinc, fruits and vegetables, and the Mediterranean diet. Nutrients may impact development of asthma through immune modulation or the child's intestinal microbiome. In spite of, or possibly because of, recommendations for early life avoidance of specific 'highly allergenic' foods including peanut in the 1990s from many national expert organizations (e.g. Canadian and British Pediatric Societies, American Academy of Pediatrics) there has been an explosion of food allergy, particularly to peanut in most high income countries (Miles and Buttriss, Nutrition Bulletin 2010). Intriguingly, studies have shown a very low prevalence of peanut allergy in Israel where peanut is commonly introduced in the first year of life compared with England where it is seldom introduced before the first birthday. This study accounted for a general heritable risk using children from a similar background (Ashkenazi Jewish) in both countries. (DuToit et al, JACI 2008). In the Danish National Birth Cohort maternal peanut (RR: 0.66; 95% CI: 0.44-0.98) and tree nut (RR: 0.83; 95% CI: 0.70-1.00) intake during pregnancy was associated with decreased risk of asthma in the child at 18 months of age. Intriguingly, there was no comment on the development of allergy in this cohort. The data being collected in the CHILD Study will allow the investigators to examine the link between maternal intake of specific foods such as peanut and the outcome of allergy to that food in the infant.
2. Low serum 25-hydroxyvitamin D values in infancy are associated with development of early childhood wheezing. Most, but not all, studies have demonstrated a relationship of maternal vitamin D insufficiency with wheezing in pre-school children. A meta-analysis of four large cohort studies found that high maternal vitamin D intake during pregnancy was protective against wheeze in children. However, a recent publication from the ALSPAC cohort shows an association of increased wheeze with increased vitamin D levels. One issue may well be polymorphisms of the Vitamin D receptor in the mother (associated with vitamin D levels during pregnancy) and in their offspring during the few years of life. The data obtained in the CHILD Study will provide the opportunity to confirm or negate the associations between levels of vitamin D and wheezing syndromes in early childhood.
3. Sensitization to cow's milk, egg or peanut, together or separately, at 1 year is a major risk factor for wheezing episodes in early infancy. Sensitization to foods has been associated with an increased risk for asthma (Rhodes et al, J Allergy Clin Immunol. 2001;108:720-5 and has recently been included in a modified Asthma Predictive Index (mAPI) (NEJM 2006;354:1985-97). The mAPI and an m2API have been validated in a small cohort as good predictors for persistent asthma at school age (Chang T et al, J Allergy Clin Immunol: In Practice 2013; 1:152-156). As yet unpublished data from a Canadian cohort show a substantial increased risk (OR 8-10) of persistent asthma in children with sensitization to a food in the first year of life (verbal communication, Becker A). The investigators will be able, using CHILD Study data, to examine these early life sensitization patterns in relation to the occurrence of wheezing episodes, and not only determine immediate relationships but also follow the children for several years to validate (or not) the Asthma Predictive Index.
4. Exposures to oxidizing agents in the prenatal period and during the first 3 months of life influence the development of atopy and wheeze at 1 year. Infants raised in Canada spend a large majority of time indoors at home. Multiple indoor air exposures have been associated with wheeze and asthma, environmental tobacco smoke (ETS) being the most widely recognized. Oxides of nitrogen, associated with gas cooking and heating, are linked with worsening asthma. Innate immune inflammatory response can be activated by common indoor exposures, including trichloramines, aldehydes (e.g., formaldehyde) and other volatile organic compounds (VOCs) in home furnishings and cleaning products.

Recent studies suggest that early-life exposure to ambient air pollution may also contribute to the development of asthma, with traffic-related air pollution (TRAP) likely playing an important role. TRAP represents a complex mixture of pollutants (particulate matter, nitrogen oxides, carbon monoxide, organic compounds) in concentrations that are variable over short distances, but that also build-up over parts of the city contributing to a variable urban background. Respiratory health risks are generally highest among those living close to busy roads with significant truck traffic, but concentration variations across urban areas have also been associated with incident asthma. The effects of TRAP on airways disease likely also depend on poorly understood interactions with a range of endogenous or exogenous factors such as genetics, co-exposures such as allergens and environmental tobacco smoke, and psychosocial stress. The CHILD Study provides an opportunity to study TRAP in four major cities with highly variable and well-characterized concentrations, and to examine relationships between TRAP, indoor air contaminants, and development of wheeze and atopy in early childhood with the intent of following these children through childhood to determine asthma outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 years and older (19 in Vancouver) 2. Residence in reasonable proximity to the delivery hospital 3. Able to read, write, and speak English 4. Willing to provide informed consent 5. Willing to consent to cord blood collection for the study 6. Planning to give birth at a designated recruitment centre participating hospital 7. Infants born at or after 35 weeks 8. Able to provide address and telephone number and names and telephone numbers of two alternate contact individuals

Exclusion Criteria:

1. Children with major congenital abnormalities or respiratory distress syndrome (RDS)
2. Expectation of moving away from a recruitment area within year 1
3. Children of multiple births
4. Children resulting from in vitro fertilization
5. Children who will not spend at least 80% of nights in the index home

Ages: 1 Day to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The 500 children in Project 500 will be representative of our full cohort. Study members have been recruited from a general population (i.e., not high-risk for asthma and allergy as are many cohorts) from recruitment bases in Vancouver, Edmonton, Winnipeg (including a rural site in Manitoba) and Toronto.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2008-08-31 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Allergic sensitization at 1 year | March 2018
  Skin prick tests to food and inhalant allergies

SECONDARY OUTCOMES:
Early childhood wheeze | Birth to one year
  Parental report of childhood wheezing
Atopic Dermatitis | Birth to one year
  Parental report of skin rashes

OTHER OUTCOMES:
Food Allergy | Birth to one year
  Parental report of food allergy

CONTACTS AND LOCATIONS:
Overall Officials: Padmaja Subbarao, MD, Study Director — University of Toronto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takaro TK, Scott JA, Allen RW, Anand SS, Becker AB, Befus AD, Brauer M, Duncan J, Lefebvre DL, Lou W, Mandhane PJ, McLean KE, Miller G, Sbihi H, Shu H, Subbarao P, Turvey SE, Wheeler AJ, Zeng L, Sears MR, Brook JR; CHILD study investigators. The Canadian Healthy Infant Longitudinal Development (CHILD) birth cohort study: assessment of environmental exposures. J Expo Sci Environ Epidemiol. 2015 Nov-Dec;25(6):580-92. doi: 10.1038/jes.2015.7. Epub 2015 Mar 25. PMID 25805254
- [Background] Moraes TJ, Lefebvre DL, Chooniedass R, Becker AB, Brook JR, Denburg J, HayGlass KT, Hegele RG, Kollmann TR, Macri J, Mandhane PJ, Scott JA, Subbarao P, Takaro TK, Turvey SE, Duncan JD, Sears MR, Befus AD; CHILD Study Investigators. The Canadian healthy infant longitudinal development birth cohort study: biological samples and biobanking. Paediatr Perinat Epidemiol. 2015 Jan;29(1):84-92. doi: 10.1111/ppe.12161. Epub 2014 Nov 18. PMID 25405552
- [Background] Subbarao P, Anand SS, Becker AB, Befus AD, Brauer M, Brook JR, Denburg JA, HayGlass KT, Kobor MS, Kollmann TR, Kozyrskyj AL, Lou WY, Mandhane PJ, Miller GE, Moraes TJ, Pare PD, Scott JA, Takaro TK, Turvey SE, Duncan JM, Lefebvre DL, Sears MR; CHILD Study investigators. The Canadian Healthy Infant Longitudinal Development (CHILD) Study: examining developmental origins of allergy and asthma. Thorax. 2015 Oct;70(10):998-1000. doi: 10.1136/thoraxjnl-2015-207246. Epub 2015 Jun 11. PMID 26069286
- [Derived] Azad MB, Robertson B, Atakora F, Becker AB, Subbarao P, Moraes TJ, Mandhane PJ, Turvey SE, Lefebvre DL, Sears MR, Bode L. Human Milk Oligosaccharide Concentrations Are Associated with Multiple Fixed and Modifiable Maternal Characteristics, Environmental Factors, and Feeding Practices. J Nutr. 2018 Nov 1;148(11):1733-1742. doi: 10.1093/jn/nxy175. PMID 30247646
- See also: Overview of the CHILD Study — http://www.canadianchildstudy.ca

DOCUMENTS (1):
  • Study Protocol (2013-04-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT03225534/Prot_000.pdf